CLINICAL TRIAL: NCT06943066
Title: The Effects of Pilates Exercises on Pain, Fatigue, Endurance, and Muscle Strength in Individuals With Non-Specific Low Back Pain
Brief Title: Pilates Exercises on Pain, Fatigue, Endurance, and Muscle Strength in Non-Specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-04-06
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Low Back Pain
Keywords: exercise
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reformer Pilates (Experimental)
  Interventions: Other: Reformer Pilates
- Pilates control (Active Comparator)
  Interventions: Other: Pilates control
- online pilates (Active Comparator)
  Interventions: Other: online pilates

INTERVENTIONS:
Other: Reformer Pilates — Reformer Pilates
  Arms: Reformer Pilates
Other: Pilates control — Pilates control
  Arms: Pilates control
Other: online pilates — online pilates
  Arms: online pilates

SUMMARY:
Pilates exercises administered under the supervision of a physiotherapist on pain, endurance, and muscle strength in individuals with non-specific low back pain, and to determine which program is more beneficial and reliable.

DETAILED DESCRIPTION:
The aim of this study is to compare the effects of different types of Pilates exercises administered under the supervision of a physiotherapist on pain, endurance, and muscle strength in individuals with non-specific low back pain, and to determine which program is more beneficial and reliable.

ELIGIBILITY:
Inclusion Criteria

* Aged between 18 and 60 years
* Non-specific low back pain for more than 12 weeks
* No clear pathological diagnosis
* Physically and cognitively capable of performing the exercises
* Pain level between 3 and 7 on the Visual Analog Scale (VAS) Exclusion Criteria
* Pregnancy
* Spinal surgery in the last 6 months
* Neurological or chronic systemic diseases
* Movement restriction due to severe pain

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-04-06 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 12 weeks
  A 10-cm line where participants mark their pain intensity, ranging from 'no pain' to 'worst pain'.
Oswestry Disability Index | 12 weeks
  A 10-section questionnaire evaluating the impact of back pain on daily activities. maximum point 56
Fatigue Severity Scale | 12 weeks
  A 9-item self-report scale where participants rate how fatigue affects their daily life on a 1-7 scale.
Heart Rate Variability | 12 weeks
  Measured using the Polar H10 sensor to evaluate autonomic nervous system activity during rest and activity.
Trunk Flexor and Extensor Endurance Tests: | 12 weeks
  Time-based static hold tests assessing core stabilization ability in flexion and extension positions.
Plank Test | 12 weeks
  Participant holds a forearm plank position, and the time until fatigue or form loss is recorded to assess core endurance.

CONTACTS AND LOCATIONS:
Locations (1):
- Hazal GENÇ, Istanbul, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No